CLINICAL TRIAL: NCT07355517
Title: Guided Biofilm Therapy Versus Conventional Ultrasonic Debridement and Polishing for the Treatment of Gingivitis in Patients With Fixed Orthodontic Appliances: A Split-Mouth Randomized Controlled Clinical Trial
Brief Title: Guided Biofilm Therapy Compared to Traditional Cleaning for Treating Gingival Inflammation in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other); Deanship of Scientific Research/Jordan University of Science and Technology (Unknown)
Responsible Party: Principal Investigator, Reem Abdel-Hafez, Associate Professor of Periodontology, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/80
Record Dates: First submitted 2025-06-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Gingivitis and Periodontal Diseases; Gingivitis; Chronic; Gingivitis; Gingival Bleeding; Periodontal Health; Gingival Health
Keywords: Gingivitis; Dental plaque; Oral hygiene; Periodontal health; Orthodontic appliances; Guided Biofilm Therapy; Scaling; Dental polishing; Scaling and polishing; Biofilm removal; Patient satisfaction; Treatment time; Clinical trial; Tooth cleaning; Non-surgical periodontal therapy; Preventive dentistry; Dental prophylaxis; Randomized controlled trial; Gingiva; Periodontium
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Bronchiolitis Obliterans Syndrome; Gingival Hemorrhage; Dental Plaque; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This study is conduct in a split mouth fashion, meaning each patient mouth is divided into halves, each half is then randomized to either the test or the control group. Therefore, the study is parallel deisgn, with one arm containing all the halves in the treatment group and the other arm containing the other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test: Guided Biofilm Therapy (Experimental): Treatment by Guided Biofilm Therapy (GBT). GBT treatment consists of supragingival and submarginal air polishing (Air-Flow Master Piezon®, EMS) with erythritol + chlorhexidine powder (PLUS®, EMS), followed by site-specific removal of calculus with ultrasonic piezoelectric scaler (Air-Flow Master Piezon®, EMS).
  Interventions: Device: Guided Biofilm Therapy
- Control: Tradition Ultrasnoic Scaling + Polishing (Active Comparator): Traditional ultrasonic debridement followed by polishing with a bristle brush and prophylactic paste.
  Interventions: Device: Traditional Ultrasonic Scaling + Polishing

INTERVENTIONS:
Device: Guided Biofilm Therapy — Guided Biofilm Therapy (GBT) focuses on the detection and targeted removal of dental biofilm. It was developed by EMS (Electro Medical Systems) and is claimed to be minimally invasive, gentle, and highly effective for both patients and practitioners.
  Key Features of GBT:
  Biofilm Detection: Uses disclosing agents to stain biofilm, making it visible for complete and accurate removal.
  Air Polishing (AIRFLOW®): A gentle, high-precision spray of air, water, and erythritol (or glycine) powder removes the biofilm.
  Subgingival Cleaning (PERIOFLOW®): Targets biofilm below the gingival margin and in periodontal pockets using a flexible nozzle and fine powder.
  Ultrasonic Debridement (PIEZON® NO PAIN): Removes remaining hard calculus with a piezoelectric scaler.
  Arms: Test: Guided Biofilm Therapy
Device: Traditional Ultrasonic Scaling + Polishing — Traditional ultrasonic scaling and polishing is a nonsurgical periodontal debridement procedure that utilizes an ultrasonic scaler-typically magnetostrictive or piezoelectric-to mechanically disrupt and remove dental calculus, dental plaque biofilm, and extrinsic stains. The procedure is followed by polishing using a bristle brush and prophylactic paste containing abrasive agents to remove extrinsic stains smooth enamel surfaces, reducing bacterial adhesion and improving esthetics. It is commonly performed as part of routine periodontal maintenance to prevent gingivitis and the progression of periodontitis.
  Other Names: Traditional Non-surgical Periodontal Debridement and Polishing; Traditional Non-surgical Periodontal Debridement and Prophylaxis
  Arms: Control: Tradition Ultrasnoic Scaling + Polishing

SUMMARY:
Why is this study being done?

This study is for people with braces who have gum inflammation (gingivitis), which is when gums are swollen and bleed easily. Braces can make it harder to clean teeth, leading to a build-up of plaque (a sticky layer of germs).

The goal is to compare two different professional dental cleaning methods to see which one works better for people with braces.

What is the main question the study is trying to answer?

The main questions are:

Which cleaning method is better at removing plaque?

Which method leads to healthier gums (less bleeding and inflammation) after 2 weeks and 8 weeks?

The study will also look at:

How long each cleaning takes.

How comfortable or uncomfortable each method is for the participant.

Which method participants like better.

What methods are being compared?

Researchers will compare two methods:

Guided Biofilm Therapy (GBT): A newer method that uses a special powder with air to remove plaque, followed by a specific ultrasonic tool to remove any hard buildup.

Conventional Cleaning: The traditional method that uses an ultrasonic tool to clean the teeth, followed by polishing with a brush and paste.

How will the study work?

This is a "split-mouth" study. This means each participant will get both cleaning methods in one visit:

One side of the mouth will get the GBT cleaning.

The other side of the mouth will get the conventional cleaning.

The side that gets each treatment is chosen by chance (randomly). This lets researchers make a very fair comparison for each person.

Who can join this study?

Participants who:

Are between 18 and 40 years old.

Have braces on both their upper and lower teeth.

Have signs of gum inflammation (gingivitis).

Are in good general health and do not smoke.

Who cannot join this study?

Participants who:

Have severe gum disease (periodontitis).

Are pregnant or breastfeeding.

Are allergic to the cleaning materials (like erythritol or chlorhexidine).

Have had a professional gum treatment in the last 3 months.

What will participants be asked to do?

If you join this study, you will be asked to:

Come in for a first visit to check your gum health.

Receive both cleaning treatments (one on each side of your mouth) during the same visit.

Answer a short questionnaire after the cleaning about your comfort and which method you preferred.

Return for two follow-up checkups (at 2 weeks and 8 weeks) so researchers can check your gum health.

DETAILED DESCRIPTION:
This randomized split-mouth controlled clinical trial is designed to assess the comparative effectiveness of Guided Biofilm Therapy (GBT) and conventional ultrasonic debridement with bristle brush polishing in patients with fixed orthodontic appliances. The trial specifically evaluates the reduction of dental plaque accumulation, gingival inflammation, treatment duration, potential adverse effects, and patient-reported outcomes such as comfort and satisfaction.

Conventional treatment will consist of full-mouth ultrasonic debridement performed with a piezoelectric scaler (frequency range 28-32 kHz, standard tip for supra- and subgingival instrumentation), followed by polishing with a nylon bristle brush mounted on a low-speed handpiece and prophylactic paste. GBT will be performed according to the standardized EMS protocol. Supragingival and subgingival air-polishing will be conducted using erythritol + 0.3% chlorhexidine powder (PLUS®, EMS, particle size <14 µm) delivered by the Air-Flow Master Piezon® device. Site-specific calculus removal will then be performed using piezoelectric instrumentation with slim tips designed for subgingival access.

At baseline, plaque disclosure will be performed using EIMS-DV 158 biofilm disclosing agents, followed by digital photographs to document biofilm distribution. Clinical indices will include plaque accumulation recorded using the Rustogi Modified Navy Plaque Index (RMNPI) and the Modified O'Leary Index, gingival inflammation assessed by the Löe and Silness Gingival Index, and bleeding on probing (BoP) recorded dichotomously at six sites per tooth. Randomization will assign one side of the mouth to GBT and the contralateral side to conventional treatment. Each treatment session will be timed using a digital stopwatch, with plaque removal endpoints recorded. Any additional instrumentation required to achieve complete plaque removal will be documented.

All clinical procedures will be performed by calibrated periodontists. Calibration will be achieved by duplicate assessment of at least 10 patients not included in the trial until intra- and inter-examiner reliability reach a kappa value of ≥0.80 for all indices. Standardized instruments and consumables will be used throughout the study to minimize variability.

Following the professional intervention, participants will receive standardized oral hygiene instructions that include the use of a soft manual toothbrush (soft bristle, end-rounded filaments) and interdental brushes selected according to embrasure size. A structured questionnaire will be administered immediately after treatment to assess perceived pain or discomfort, treatment tolerability, perceived oral cleanliness, and preference between the two modalities using a validated 5-point Likert scale.

Clinical re-evaluations will be performed at 2 weeks and 8 weeks. The same indices (plaque, gingival inflammation, BoP) will be reassessed by calibrated examiners. Oral hygiene instructions will be reinforced at each visit.

The trial will be conducted in accordance with the Declaration of Helsinki (2013) and Good Clinical Practice (GCP) guidelines. Approval has been granted by the Institutional Review Board (IRB) of Jordan University of Science and Technology. Written informed consent will be obtained from all participants prior to enrollment. Adverse events will be documented, monitored, and reported according to IRB requirements.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* Presence of fixed orthodontic appliances in both upper and lower arches for at least 1 month
* Diagnosed with generalized biofilm-induced gingivitis (defined as Bleeding on Probing (BoP) > 30% of sites)
* Presence of a minimum of 10 teeth per side
* Systemically healthy
* Non-smoker
* Motivated and able to maintain good oral hygiene
* Willing and able to provide written informed consent

Exclusion Criteria:

* Diagnosed with periodontitis or a history of periodontitis
* Pregnant or lactating women
* Allergy to erythritol or chlorhexidine
* Presence of dental caries or overhanging restorations
* Presence of more than 6 teeth with gingival enlargement grade II or III according to the Angelopoulos and Goaz Index
* Received periodontal treatment within the last 3 months
* Expected to complete orthodontic treatment before the end of the study
* Unwillingness to undergo the proposed treatment or follow-up visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
Change in Rustogi Modified Navy Plaque Index (RMNPI) | Baseline, 2 weeks, 8 weeks
  The RMNPI is a detailed plaque scoring system that evaluates the buccal/labial surfaces of teeth by dividing each surface into nine distinct areas. Each area is scored dichotomously as 1 (plaque present) or 0 (plaque absent). In this study, due to the presence of orthodontic brackets, only four surfaces (mesial, distal, incisal, and gingival) will be evaluated, modifying the total number of assessed sections. The index is sensitive to small areas of plaque accumulation and provides data on incisal, gingival, and interproximal plaque levels. A plaque disclosing agent will be used prior to scoring. The Modified O'Leary Index will be used on lingual/palatal surfaces.
Change in Bleeding on Probing Percentage (BoP%) | Baseline, 2 weeks, 8 weeks
  BoP will be recorded dichotomously at six sites per tooth, and BoP% will be calculated as the percentage of bleeding sites relative to total measured sites.

SECONDARY OUTCOMES:
Change in Gingival Index (GI) | Baseline, 2 weeks, 8 weeks
  The Gingival Index by Löe and Silness measures gingival inflammation based on color, consistency, and bleeding on probing. Scoring is as follows:
  0 = Normal gingiva
  1. = Mild inflammation (slight change in color, slight edema, no bleeding on probing)
  2. = Moderate inflammation (redness, edema, glazing, bleeding on probing)
  3. = Severe inflammation (marked redness and edema, ulceration, spontaneous bleeding)
Change in Probing Depth (PD) | Baseline, 2 weeks, 8 weeks
  Periodontal probing depth will be measured at six points per tooth using a calibrated periodontal probe. The distance (in mm) from the gingival margin to the base of the periodontal pocket will be recorded.
Change in Plaque Index (Löe and Silness) | Baseline, 2 weeks, 8 weeks
  The Löe and Silness Plaque Index evaluates the thickness of plaque at the gingival margin of the tooth. It is scored on a scale from 0 to 3:
  0 = No plaque
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth, visible only by disclosing solution or by running a probe across the surface
  2. = Moderate accumulation of soft deposits visible to the naked eye
  3. = Abundance of soft matter This index will be used on the lingual/palatal surfaces of teeth using disclosing agents.

OTHER OUTCOMES:
Total Treatment Time Per Side | Day 1, postoperative
  The time (in minutes) required to complete the debridement procedure per side (traditional or GBT) will be measured. Time starts at the beginning of treatment and ends when the clinician is satisfied with plaque removal. Additional time required to remove residual plaque (as shown by reapplication of disclosing agent) will be recorded separately.
Patient-Reported Pain/Discomfort Level | Immediately post-treatment
  Patients will report discomfort or pain experienced during each treatment using a 5-point Likert scale:
  1. = No discomfort
  2. = Mild
  3. = Moderate
  4. = Considerable
  5. = Severe
Patient-Reported Feeling of Cleanliness | Immediately post-treatment
  Patients will indicate how clean their teeth feel after treatment using a 5-point Likert scale (1 = not clean at all, 5 = very clean).
Patient Preference Between the Two Treatment Modalities | Immediately post-treatment
  Patients will be asked which of the two treatment modalities (Guided Biofilm Therapy [GBT] or traditional ultrasonic debridement with polishing) they preferred, patients will only choose 1 of the two as their preferred method

CONTACTS AND LOCATIONS:
Overall Officials: Reem Abdel-Hafez, Doctor of Clinical Dentistry, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) including demographics, primary and secondary outcome measures, and adverse events. Data will be made available beginning 12 months after publication of the primary results, and will be accessible to qualified researchers upon reasonable request, subject to data-sharing agreements and IRB approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after publication of primary results and will remain available for 5 years via a controlled access repository upon request and data use agreement.
Access Criteria: Qualified researchers affiliated with academic institutions, healthcare organizations, or nonprofit research centers will be able to request access to the de-identified individual participant data (IPD) and supporting documents, including the Study Protocol, Statistical Analysis Plan (SAP), and Analytic Code.
  Requests for access will be reviewed by the study sponsor or data access committee to ensure appropriate use and ethical standards.
  Approved users will receive access via a secure online data repository, after signing a data use agreement that outlines terms of use, privacy protections, and publication rights.